CLINICAL TRIAL: NCT07228988
Title: Patient-Related Outcomes of Digital and Conventional Removable Partial Dentures..A Crossover Randomised Clinical Trial
Brief Title: Comparison of Patient Satisfaction Between Conventional and Digital Removable Partial Dentures
Acronym: TRI-RBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Enas Mesallum, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 209-12-24 ethical approval
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Partially Edentulous Patients
Keywords: Removable partial denture; Patient satisfaction; Digital partial denture; PEEK; 3D printed printed denture; Oral health quality of life
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: 3 intervention arms will be used as participants are randomly assigned to one of the 3 dentures Conventional, 3D printed, or PEEK for one month then after one week washout every patient will switch to another type of dentures for another one month, the final phase after a week of rest each patient will try the third type
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional cast Co-Cr removable partial denture (Active Comparator): This type of RPD is constructed from Cobalt Chromium metal framework using the lost wax technique conventional casting of a wax pattern made on an investment cast.. Each participant used the conventional denture for 30 days then they received the VAS and OHIP-14 questionnaire about their denture experience..Then wait one week without any dentures until they received the second denture type
  Interventions: Device: Conventional cast Cr-Co RPDs
- 3D Printed Cr-Co removable partial denture (Experimental): This is a digital RPD made from Cobalt Chromium metal which is printed by a 3D printer using selective laser melting technique..Each participant used the 3D printed denture for 30 days then they received the VAS and OHIP-14 questionnaire about their denture experience..Then wait one week without any dentures until they received the next denture type
  Interventions: Device: 3D Printed Cr-Co RPDS
- Milled PEEK removable partial dentures (Experimental): This is a digital type of RPD made by milling polyetheretherktone discs using a milling machine..Each participant used the PEEK denture for 30 days then they received the VAS and OHIP-14 questionnaire about their denture experience..Then wait one week without any dentures until they received the other denture type
  Interventions: Device: Milled PEEK RPDs

INTERVENTIONS:
Device: Conventional cast Cr-Co RPDs — Conventional Cr-Co RPD is constructed by the standard lost wax technique to act as active comparator being the traditional way of RPD construction
  Arms: Conventional cast Co-Cr removable partial denture
Device: 3D Printed Cr-Co RPDS — 3D Printed Cr-Co was constructed digitally using Laser Melting technology to 3D print the Cr-Co RPD to the same design used with the conventional and the patient used every denture for 30 days with one week wash out
  Arms: 3D Printed Cr-Co removable partial denture
Device: Milled PEEK RPDs — PEEK disc was milled using milling machine to construct RPD framework to the same design as other 2 groups, each patient will use all the 3 dentures for one month but with different sequences, after each type one week washout separated between the groups
  Arms: Milled PEEK removable partial dentures

SUMMARY:
Study type: cross over within subject clinical trial Primary aim: To compare patient satisfaction among three different RPDs: conventional cast Co-Cr, 3D-printed Co-Cr, and PEEK RPDs.

Secondary aim: To evaluate the impact of these RPDs on oral health-related quality of life and patient preference among these RPDs

DETAILED DESCRIPTION:
A within-subject randomized crossover clinical was conducted at the Faculty of Dentistry, King Abdulaziz University after obtaining an ethical approvalfrom the Faculty Ethical Committee. All patients have signed a consent before being enrolled in the study.

Each participant received three RPDs using three manufacturing techniques (conventional cast Co-Cr, 3D-printed Co-Cr, and milled PEEK) fabricated to the same RPD design specifications. Each RPD worn for 30 days with a one-week washout period between the trial phases.

Participants were selected from partially edentulous patients fulfilling mandibular Kennedy Class I with the first or second premolars as the last abutment teeth bilaterally . Inclusion criteria include good oral hygiene, healthy mucosa, and absence of systemic diseases affecting oral tissues. Exclusion criteria include allergy to materials, poor compliance, or history of temporomandibular disorders.

Sample size estimation is based on detecting a moderate effect size (f = 0.25) with 80% power and α = 0.05, requiring at least 30 participants. To account for possible dropouts, a total of 36 patients was recruited.

Patient satisfaction was assessed using the Visual Analogue Grade (VAG) scale (0-100 mm). The VAG evaluates satisfaction domains such as comfort, esthetics, speech, and mastication, while OHIP-14 measures the impact of oral health on quality of life through 14 questions covering 7 domains. At the end of all the treatment phases participants determined the most preferred denture by answering single choice question of the best overall denture among the three types.

Results will be statistically analysed using one ANOVA test and Tukeys test if the difference between groups is significant

ELIGIBILITY:
Inclusion Criteria:

- Partially edentulous patients with mandibular Kennedy class I, last abutment is the first or second premolars, maxillary arch is dentate or restored, good oral hygiene

Exclusion Criteria:

* Any systemic diseases that affect oral health, periodontal disease, improper patient compliance, TMD

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction using VAG | Delivery of the first denture type 1st questionnaire 30 days after receiving the first denture 7 days wash out Delivery of the second denture type 2nd questionnaire 30 days after using the denture 7 days wash out Final questionnaire after 30 days
  Visual Analogue Grade 100 mm scale is used to measure patient satisfaction and comfort as zero indicates the worst and 100 indicates the best response

SECONDARY OUTCOMES:
Oral Health related Quality of Life OHRQoL | Delivery of the first denture type 1st questionnaire 30 days after receiving the first denture 7 days wash out Delivery of the second denture type 2nd questionnaire 30 days after using the denture 7 days wash out Final questionnaire after 30 days
  OHIP-14 questionnaire is used to assess the OHRQol
Patient preference | After all the three dentures treatment phase 30 days after the delivery of the last denture according to sequence randomisation Study time line was 6 months from recruitment to final questionnaire
  Single short end question to select one type of denture that was preferred by the patient after using all the three types

CONTACTS AND LOCATIONS:
Overall Officials: Enas E. Mesallum, PhD, Study Director — Assistant Professor of Prosthodontics, King Abdulaziz University
Locations (2):
- Saudi Arabia (2):
  - Faulty of dentistry King Adbulaziz University-KAU, Jeddah, Western
  - King Adbulaziz University-KAU, Jeddah, Westren

IPD SHARING:
Plan to Share IPD: No
Only summary statistics will be included in the published article later on

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT07228988/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT07228988/ICF_001.pdf